CLINICAL TRIAL: NCT04925024
Title: Evaluation of Lomecel-B™ Injection in Patients With Hypoplastic Left Heart Syndrome (HLHS) : A Phase IIb Clinical Trial.
Brief Title: Evaluation of Lomecel-B™ Injection in Patients With Hypoplastic Left Heart Syndrome (HLHS): A Phase IIb Clinical Trial.
Acronym: ELPIS II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Ann & Robert H Lurie Children's Hospital of Chicago (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-4531; 7UG3HL148318-02 (NIH); 1U24HL148316-01A1 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; Pediatrics; Heart Defects; Congenital Cardiovascular Diseases; Stem Cells
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lomecel B Group (Experimental): Participants randomized to receive Lomecel-B injections during their Stage II palliation.
  Interventions: Biological: Lomecel-B medicinal signaling cells
- No Study Intervention Control Group (No Intervention): Participants randomized to receive no study intervention during their Stage II palliation.

INTERVENTIONS:
Biological: Lomecel-B medicinal signaling cells — A single administration of Lomecel-B will be performed via 6-10 intramyocardial injections into the right ventricle during the participant's standard of care stage II palliation. Dosing is based on body weight. Each patient will be given 2.5 x 10^5 cells per kg of body weight. The entire dose of the cells will be roughly 600 microliters.
  Arms: Lomecel B Group

SUMMARY:
The purpose of this study is to test whether Lomecel-B™ works in treating patients with hypoplastic left heart syndrome (HLHS) and to gather additional information about the safety of Lomecel-B. Lomecel-B contains human mesenchymal stem cells (MSCs) as the active ingredient. MSCs are special cells in the body that are able to change into other types of cells, such as heart, blood, and muscle cells. MSCs are found in various tissues of the body, such as the bone marrow, which is the spongy tissue inside of your bones. Lomecel-B uses MSCs from bone marrow of unrelated young healthy donors. These are called "allogeneic", and do not require donor matching to the patient.

ELIGIBILITY:
Inclusion:

All participants must have HLHS (includes all types) requiring Stage II palliation (Glenn or Hemi-Fontan operation).

Exclusion:

1. Requirement for ongoing mechanical circulatory support immediately prior to Stage II palliation within 5 days
2. Need for concomitant surgery for aortic coarctation or tricuspid valve repair or Endocardial fibroelastosis (EFE) resection or left ventricle recruitment procedures
3. Undergoing the Stage I (Norwood) procedure that does not have HLHS
4. Serum positivity for: human immunodeficiency virus (HIV); hepatitis B virus surface antigen (HBV BsAg); and/or viremic hepatitis C virus (HCV). This criterion can be ascertained by one of three ways:

   1. Documented history of mother's testing conducted during pregnancy
   2. Documented history of participants testing.
   3. If above documentation is not available blood will be obtained from participant at Screening/Baseline.
5. Parent/guardian that is unwilling or unable to comply with necessary follow-up
6. Unsuitability for the study based on the Investigator's clinical opinion
7. Known hypersensitivity to dimethyl sulfoxide (DMSO)
8. Presence of a pacemaker, or anticipated placement of a pacemaker, at the time of the Stage II palliation

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in right ventricular ejection fraction (RVEF) | Baseline, 12 Months
  Efficacy will be reported as change in right ventricular ejection fraction (RVEF) assessed as a percentage and will be measured via cardiac magnetic resonance (CMR) imaging.

SECONDARY OUTCOMES:
Change in right ventricular ejection fraction (RVEF) | Baseline, 6 Months
  Efficacy will be reported as change in right ventricular ejection fraction (RVEF) assessed as a percentage and will be measured via cardiac magnetic resonance (CMR) imaging.
Change in right ventricular mass index at diastole | Baseline, 12 Months
  Efficacy will be reported as change in right ventricular mass index at diastole assessed as g/m^2 and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in right ventricular end-diastolic volume index (RVEDVI) | Baseline, 12 Months
  Efficacy will be reported as change in right ventricular end diastolic volume index (RVEDVI) assessed as ml/m^2 and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in right ventricular end-systolic volume index (RVESVI) | Baseline, 12 Months
  Efficacy will be reported as change in right ventricular end systolic volume index (RVESVI) assessed as ml/m^2 and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in right ventricular global longitudinal strain and strain rate | Baseline, 12 Months
  Efficacy will be reported as change in right ventricular global longitudinal strain and strain rate assessed as % and s^-1 respectively and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in right ventricular global circumferential strain and strain rate | Baseline, 12 Months
  Efficacy will be reported as the change in right ventricular global circumferential strain and strain rate as % and s^-1 respectively, and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in right atrial volume index | Baseline, 12 Months
  Efficacy will be reported as the change in right atrial volume index as ml/m^2 and will be measured via serial cardiac magnetic resonance (CMR) imaging.
Change in tricuspid regurgitation severity | Baseline, 12 Months
  Efficacy will be reported as change in the categorical qualitative assessment of tricuspid valve regurgitation (trivial, mild, moderate, severe) and will be measured via transthoracic echocardiography.
Change in weight | Baseline, 12 Months
  Efficacy measured as change in participant's weight in kg and will be measured serially to assess change in somatic growth.
Change in length (height) | Baseline, 12 Months
  Efficacy measured as change in participant's length (height) in cm and will be measured serially to assess change in somatic growth.
Change in head circumference | Baseline, 12 Months
  Efficacy measured as change in participant's head circumference in cm and will be measured serially to assess change in somatic growth.
Change in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) | Baseline, 12 Months
  Efficacy measured as change in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) in pg/ml and will be measured serially by blood draw.
Change in modified Ross Heart Failure Classification score | Baseline, 12 Months
  The Ross Heart Failure Classification provides a global assessment of heart failure severity in infants. Efficacy measured as change in classification and will be measured serially via physician's assessment using the modified Ross Heart Failure Classification; classifications defined as Class 1 (no limitations of physical activity); Class 2 (may experience symptoms during moderate exercise but not during rest); Class 3 (symptoms with minimal exertion that interfere with normal daily activity); Class 4 (unable to carry out physical activity/has symptoms at rest that worsen with exertion).
Change in PedsQL™ Infant Scales | Baseline, 12 Months
  The PedsQL™ Infant Scales is a generic health related quality of life instrument specifically for healthy and ill infants ages 1-24 months. Efficacy measured as change in PedsQL total improvement score and will be measured serially by parental proxy-report. Higher scores are indicative of better quality of life.
Freedom from unplanned catheter intervention needed to address the pulmonary arteries or aorta. | Baseline, 12 Months
  Efficacy measured as the number and percentage of participants who do not undergo unplanned catheter interventions to address pulmonary arteries or the aorta.
Change in biomarkers/cytokines | Baseline, 12 Months
  Efficacy measured as change in biomarkers/cytokines in pg/ml and/or ng/ml and will be measured serially by blood draw.
Participants experiencing treatment emergent serious adverse events (TE-SAEs) | 30 days post Stage II palliation
  Safety will be reported as the number of participants experiencing treatment emergent serious adverse events (TE-SAEs) assessed by treating physician within the 30 days following study procedure. These include: all-cause mortality; greater than 30 seconds of sustained/symptomatic ventricular tachycardia requiring intervention; cardiogenic shock; unplanned cardiovascular operation for bleeding due to right ventricular intramyocardial injection site bleeding in the first five days after stage II palliation; sepsis; need for new permanent pacemaker; stroke or embolic event to the brain
Participants experiencing major adverse cardiac events (MACE) | Baseline, 12 Months
  Safety will be reported as the number of participants with adjudicated events including worsening heart failure; listed for heart transplant; heart failure hospitalization; cardiovascular mortality

CONTACTS AND LOCATIONS:
Overall Officials: Stu Berger, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (10):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Advocate Children's Hospital, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Nebraska, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaushal S, Hare JM, Hoffman JR, Boyd RM, Ramdas KN, Pietris N, Kutty S, Tweddell JS, Husain SA, Menon SC, Lambert LM, Danford DA, Kligerman SJ, Hibino N, Korutla L, Vallabhajosyula P, Campbell MJ, Khan A, Naioti E, Yousefi K, Mehranfard D, McClain-Moss L, Oliva AA, Davis ME. Intramyocardial cell-based therapy with Lomecel-B during bidirectional cavopulmonary anastomosis for hypoplastic left heart syndrome: the ELPIS phase I trial. Eur Heart J Open. 2023 Jan 11;3(2):oead002. doi: 10.1093/ehjopen/oead002. eCollection 2023 Mar. PMID 36950450
- See also: ELPIS II study website — http://www.elpistrial.org
- See also: Earlier phase I study (ELPIS) — https://clinicaltrials.gov/ct2/show/NCT03525418